CLINICAL TRIAL: NCT04319757
Title: A Phase I, Open Label, Dose Escalation Study of ACE1702 Cell Immunotherapy in Subjects With Advanced or Metastatic HER2-expressing Solid Tumors
Brief Title: ACE1702 in Subjects With Advanced or Metastatic HER2-expressing Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acepodia Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE1702-001
Record Dates: First submitted 2020-03-18; First posted 2020-03-24 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced Solid Tumor; Metastatic Cancer; Solid Tumor; HER2-positive Gastric Cancer; HER2-positive Metastatic Breast Cancer
Keywords: NK Cell Therapy; Cellular Therapy; Breast Cancer; Gastric Cancer; Ovarian Cancer; Endometrial Cancer; Metastatic Cancer; Colorectal Cancer; Head and Neck Cancer; Pancreatic Cancer; Bladder Cancer; Non-small-cell Lung Carcinoma
MeSH Terms: conditions — Neoplasm Metastasis; Breast Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Pancreatic Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ACE1702 Dose Level 1 (Experimental): Lympho-conditioning agents followed by ACE1702 (anti-HER2 oNK cells) will be administered to patients with advanced or metastatic, HER2-expressing solid tumors. HER2 expressing is defined has having HER2 immunohistochemistry (IHC) 2+ or above.
  Dose Level: 1 Planned number of subjects: 1 to 6
  Interventions: Drug: ACE1702; Drug: Cyclophosphamide; Drug: Fludarabine
- ACE1702 Dose Level 2 (Experimental): Lympho-conditioning agents followed by ACE1702 (anti-HER2 oNK cells) will be administered to patients with advanced or metastatic, HER2-expressing solid tumors. HER2 expressing is defined has having HER2 IHC 2+ or above.
  Dose Level: 2 Planned number of subjects: 1 to 6
  Interventions: Drug: ACE1702; Drug: Cyclophosphamide; Drug: Fludarabine
- ACE1702 Dose Level 3 (Experimental): Lympho-conditioning agents followed by ACE1702 (anti-HER2 oNK cells) will be administered to patients with advanced or metastatic, HER2-expressing solid tumors. HER2 expressing is defined has having HER2 IHC 2+ or above.
  Dose Level: 3 Planned number of subjects: 3 to 6
  Interventions: Drug: ACE1702; Drug: Cyclophosphamide; Drug: Fludarabine
- ACE1702 Dose Level 4 (Experimental): Lympho-conditioning agents followed by ACE1702 (anti-HER2 oNK cells) will be administered to patients with advanced or metastatic, HER2-expressing solid tumors. HER2 expressing is defined has having HER2 IHC 2+ or above.
  Dose Level: 4 Planned number of subjects: 3 to 6
  Interventions: Drug: ACE1702; Drug: Cyclophosphamide; Drug: Fludarabine
- ACE1702 Dose Level 5 (Experimental): Lympho-conditioning agents followed by ACE1702 (anti-HER2 oNK cells) will be administered to patients with advanced or metastatic, HER2-expressing solid tumors. HER2 expressing is defined has having HER2 IHC 2+ or above.
  Dose Level: 5 Planned number of subjects: 3 to 6
  Interventions: Drug: ACE1702; Drug: Cyclophosphamide; Drug: Fludarabine
- ACE1702 Dose 6 (Experimental): Lympho-conditioning agents followed by ACE1702 (anti-HER2 oNK cells) will be administered to patients with advanced or metastatic, HER2-expressing solid tumors. HER2 expressing is defined has having HER2 IHC 2+ or above.
  Dose Level: 6 Planned number of subjects: 3 to 6
  Interventions: Drug: ACE1702; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: ACE1702 — ACE1702 cellular therapy (anti-HER2 oNK cells) given intravenously
Drug: Cyclophosphamide — Lympho-conditioning agent
Drug: Fludarabine — Lympho-conditioning agent

SUMMARY:
ACE1702 (anti-HER2 oNK cells) is an off-the-shelf Natural Killer (NK) cell product that targets human HER2-expressing solid tumors. The ACE1702-001 phase I study aims to evaluate the safety and tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of ACE1702 in patients with advanced or metastatic HER2-expressing tumors, and to determine the phase Ib/II starting dose for ACE1702.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Subjects must be ≥ 18 years of age ( ≥ 20 years of age for Taiwan site)
* Subject with advanced or metastatic solid tumors that is not amenable to surgical resection and is not eligible or has refused other approved therapeutic options that have demonstrated clinical benefit.
* Histologically confirmed HER2 expression.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1
* Measurable or non-measurable evaluable disease according to RECIST 1.1
* Adequate hematologic and end-organ function at baseline
* Oxygen saturation via pulse oxygenation ≥ 90% at rest on room air

Exclusion Criteria:

* Untreated central nervous system (CNS) metastases
* Multiple primary malignancies
* Clinically significant cardiovascular disease such as New York Heart Association (NYHA) cardiac disease (class III or greater)
* Pregnant or lactating female
* Serious, uncontrolled medical disorder that, in the opinion of the Investigator, would impair the ability of the subject to receive study treatment
* History of autoimmune or immune mediated symptomatic disease
* Any anti-cancer chemotherapy or targeted small molecule therapy, or experimental therapy/device within 4 weeks or 5 half-lives of the drug prior to planned start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Adverse events, including Dose Limiting Toxicities (DLTs) and Serious Adverse Events (SAEs) | Day 7 through Day 28 / Day 4 through Day 25
  Number of subjects experiencing adverse events, and the frequency and severity of adverse events.
  Endpoint for determining the Maximum Tolerated Dose (MTD). If MTD is not identified, the highest dose administered becomes the Maximum Administered Dose (MAD).
Phase Ib/II starting dose for ACE1702 | Through study completion, up to 1 year
  The recommended phase Ib/II starting dose based on MTD. If MTD is not reached, then the recommended phase Ib/II dose will be determined based on the MAD, safety data, and pharmacodynamics data.

SECONDARY OUTCOMES:
Quantify NK cell persistence after administering ACE1702 | Day 21
  Duration of ACE1702 persistence
Evaluate immune function after administering ACE1702 | Day 21
  Measurement of serum cytokine levels, pg/mL (Interferon-γ, TNF-α, IL-2, IL-6, IL-8 and IL-10) at set timepoints

OTHER OUTCOMES:
Tumor response using Response Evaluation Criteria In Solid Tumors Assessment (RECIST) version 1.1 | Day 35 (+7 day window) of each 6 week cycle, up to 24 months
  Tumor response via radiographic assessments
Shift in serum tumor marker values (CA-125, CA 19-9, and CEA levels, in applicable tumor types) | Day 35 (+7 day window) of each 6 week cycle, up to 24 months
  Tumor response via tumor marker assessments (in applicable tumor types)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, MD, Study Director — Acepodia Biotech, Inc.
Locations (3):
- United States (2):
  - Northwestern Univeristy, Chicago, Illinois
  - MD Anderson Cancer Center, Houston, Texas
- Taipei Veteran General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No